CLINICAL TRIAL: NCT01162512
Title: Telephone-Based Physical Activity Intervention in Obese Youth
Brief Title: Telephone Physical Activity Intervention in Obese Youth
Acronym: TPAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Katrina D DuBose, Associate Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECU-2010-01
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Obesity
Keywords: physical activity; obesity; adolescents; telephone; BMI; body mass index
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity (Experimental): Participants will receive 7 weeks of weekly news letters and phone calls. The news letters and phone calls will include information about physical activity and ways to increase physical activity levels. This is in addition the standard medical care.
  Interventions: Behavioral: physical activity
- Standard Medical Care (No Intervention): Participants will receive standard medical care

INTERVENTIONS:
Behavioral: physical activity — physical activity counseling sessions will occur by telephone weekly for 2 months
  Arms: Physical Activity

SUMMARY:
The purpose of this study is to examine the effectiveness of a telephone-based physical activity (PA) intervention in obese adolescents attending a Health Weight Comprehensive Clinic. Secondary aims focus on increasing the amount of change in obesity markers, namely waist circumference and BMI z-scores. The investigators hypothesize the following: 1.The telephone-based PA intervention will increase PA levels above the mail group; and 2. The telephone-based PA intervention will provide changes in waist circumference and BMI z-scores above the mail group.

DETAILED DESCRIPTION:
Obesity rates in youth have tripled over the past 20 years. Physical activity aids in weight loss and is critical for weight maintenance. Further, physical activity has other physiological and psychological benefits. Obese youth often see specialists for weight loss treatment. Treatment in a pediatric population uses a multi-component approach, but physical activity if often overlooked. Combining physical activity information with physician care and nutritional information could improve weight loss and the overall health of these obese children.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 18 years old
* attending the ECU Pediatric Comprehensive Healthy Weight Clinic

Exclusion Criteria:

* must be able to read and write in English
* must be able to participate in physical activity

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
physical activity | 4 months
  physical activity levels during the 2 month intervnetion will be measured and then physical activity will also be measured during a 2 month follow up period

SECONDARY OUTCOMES:
BMI | 4 months
  waist circumference and weight and height will be measured. BMI will be calculated. After the 2 month intervention period the amount of change in waist circumference and BMI will be quantified. These measures will also be examined after a 2 month follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Katrina D DuBose, PhD, Principal Investigator — East Carolina University; David Collier, MD, PhD, Study Chair — East Carolina University; Lesley Lutes, PhD, Study Chair — East Carolina University; Amy Gross-McMillan, PT, PhD, Study Chair — East Carolina University
Locations (1):
- ECU Pediatric Comprehensive Healthy Weight Clinic, Greenville, North Carolina, United States